CLINICAL TRIAL: NCT03598283
Title: A Prospective Study to Evaluate the Outcome of Liver, Pancreas and Thyroid Function in Severely Burned Patients
Brief Title: Liver, Pancreas and Thyroid Function in Burn Patients
Status: Withdrawn | Type: Observational
Why Stopped: The study PI has left the institution.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0053
Record Dates: First submitted 2018-06-27; First posted 2018-07-26 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Burns; Liver Fibroses; Pancreas Disease; Thyroid Diseases
MeSH Terms: conditions — Burns; Liver Cirrhosis; Pancreatic Diseases; Thyroid Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severely burned patients: In this prospective study, the extent to which severe burn injuries affect the morphology and function of liver, pancreas and thyroid. The evaluation of the liver will be performed non-invasively with liver fibrosis scores based on standard blood parameters, the ultrasound-guided measurement of the liver size and the measurement of liver stiffness (correlated with liver fibrosis) and controlled attenuation parameter (CAP, correlated with hepatic steatosis) via transient elastography (FibroScan©, Echosens SA, Paris, France). The thyroid will be assessed by ultrasound and standard blood parameters and the pancreas by standard blood parameters only, respectively.
  Interventions: Device: Ultrasound/transient elastography

INTERVENTIONS:
Device: Ultrasound/transient elastography — The evaluation of the liver will be performed non-invasively with liver fibrosis scores based on standard blood parameters, the ultrasound-guided measurement of the liver size and the measurement of liver stiffness (correlated with liver fibrosis) and controlled attenuation parameter (CAP, correlated with hepatic steatosis) via transient elastography (FibroScan©, Echosens SA, Paris, France). The thyroid will be assessed by ultrasound and standard blood parameters and the pancreas by standard blood parameters only, respectively.

SUMMARY:
The purpose of this study is to determine the extent to which severe burn injuries affect the morphology and function of liver, pancreas and thyroid. The evaluation of the liver will be performed non-invasively with liver fibrosis scores based on standard blood parameters and the measurement of liver stiffness (correlated with liver fibrosis) and controlled attenuation parameter (CAP, correlated with hepatic steatosis) via transient elastography (FibroScan©, Echosens SA, Paris, France). The thyroid and the pancreas will be assessed via ultrasound (GE Medical Systems, Waukesha, USA) and standard blood parameters, respectively.

DETAILED DESCRIPTION:
In this prospective study, the extent to which severe burn injuries affect the morphology and function of liver, pancreas and thyroid. The evaluation of the liver will be performed non-invasively with liver fibrosis scores based on standard blood parameters, the ultrasound-guided measurement of the liver size and the measurement of liver stiffness (correlated with liver fibrosis) and controlled attenuation parameter (CAP, correlated with hepatic steatosis) via transient elastography (FibroScan©, Echosens SA, Paris, France). The thyroid will be assessed by ultrasound and standard blood parameters and the pancreas by standard blood parameters only, respectively.

The patient will be enrolled during the first days on their admission to the intensive care burn unit, if they meet the inclusion criteria and no exclusion criteria are met. The first assessment of liver, pancreas and thyroid function will be performed within the first 48 hours of admission. The same measurements maybe be repeated approximately weekly until discharge, respectively. Furthermore at any follow-up visit up to 15 years post-burn if the patient consents to further participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients with partial thickness burns. Only patients who sign an IRB-approved consent (≥18 years old) or assent and have their legal guardian consenting to their participation (6 months - 17 years old) will be included.

* Patient age > 6 months
* Total body surface area (TBSA) burned ≥ 30 %
* Flame, electrical, scald or chemical injury, contact burn
* Toxic epidermal necrolysis (TENS)

Exclusion Criteria:

* Patient < 6 months
* TBSA burned < 30 %

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients older than six months
Study Population: The investigator's study population will include pediatric as well as adult patients with any type of burn injury or toxic epidermal necrolysis (TENS).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Liver stiffness (kPa) | 24 months
  Measured via transient elastography
Controlled Attenuation Parameter | 24 months
  Measured via transient elastography
Liver diameter (cm) | 24 months
  Measured via Ultrasound
Platelet count (/nl) | 24 months
  Liver function (blood tests)
High-density lipoprotein (mg/dl) | 24 months
  Liver function (blood tests)
Low-density lipoprotein (mg/dl) | 24 months
  Liver function (blood tests)
Triglycerides (mg/dl) | 24 months
  Liver function (blood tests)
Cholesterol (mg/dl) | 24 months
  Liver function (blood tests)
Alanine-aminotransferase (U/dl) | 24 months
  Liver function (blood tests)
Aspartate-aminotransferase (U/dl) | 24 months
  Liver function (blood tests)
Gamma glutamyltransferase (U/dl) | 24 months
  Liver function (blood tests)
Alkaline phosphatase (U/dl) | 24 months
  Liver function (blood tests)
Bilirubin (ng/dl) | 24 months
  Liver function (blood tests)
Albumin (g/dl) | 24 months
  Liver function (blood tests)

SECONDARY OUTCOMES:
Thyroid volume (ml) | 24 months
  Measured via Ultrasound
T3 level (ng/dl) | 24 months
  Thyroid function (blood tests)
T4 level (ng/dl) | 24 months
  Thyroid function (blood tests)
Thyroid-stimulating hormone level (U/l) | 24 months
  Thyroid function (blood tests)
Lipase (U/l) | 24 months
  Pancreas function (blood tests)
Amylase (U/l) | 24 months
  Pancreas function (blood tests)
Height (kg) | 24 months
  General patient data
Weight (kg) | 24 months
  General patient data

CONTACTS AND LOCATIONS:
Overall Officials: David N. Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- Tina Mack-Moshay, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided